CLINICAL TRIAL: NCT01732406
Title: Effect of Growth Hormone Receptor Antagonism and Somatostatin Analog Administration on Quality of Life
Brief Title: Acromegaly Treatment Quality of Life Study
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Assistant Physician in Medicine, Massachusetts General Hospital
Other Study IDs: 2012P001556
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acomegaly with Pegvisomant: Patients receiving pegvisomant monotherapy from own doctor to treat acromegaly.
- Acromegaly with somatostatin analog: Patients receiving somatostatin analog monotherapy from own doctor to treat acromegaly
- Active Acromegaly: Patients not on drugs for treatment of acromegaly

SUMMARY:
The investigators hypothesize that treatment of acromegaly will be associated with an improvement in quality of life compared to active acromegaly. At the same time, they will also be studying the effects of different acromegaly treatments on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Active acromegaly or receiving pegvisomant monotherapy or receiving somatostatin analog monotherapy

Exclusion Criteria:

* Untreated thyroid or adrenal insufficiency. Subjects on replacement therapy must be stable for at least 3 months prior to entry into the study
* Initiation or discontinuation of testosterone or estrogen within 3 months of entry
* Pregnant and nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be 3 groups/cohorts: 1) Patients with active acromegaly (n=35), 2) patients receiving pegvisomant monotherapy to treat acromegaly (n=31), and 3) patients receiving somatostatin analog monotherapy to treat acromegaly (n=60)
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acomegaly With Pegvisomant | Acromegaly With Somatostatin Analog | Active Acromegaly
Started | 31 | 60 | 35
Completed | 31 | 60 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with IGF-1 levels not consistent with assigned group were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acomegaly With Pegvisomant | Acromegaly With Somatostatin Analog | Active Acromegaly | Total
Number analyzed (Participants) | 29 | 55 | 32 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (16) | 52 (13) | 50 (15) | 51 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 34 | 17 | 72
  Male | 8 | 21 | 15 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 28 | 52 | 29 | 109
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 26 | 49 | 28 | 103
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30 (6) | 30 (7) | 30 (5) | 30 (6)
IGF-1 Level [Mean (Standard Deviation); unit: ng/ml] | 176 (58) | 174 (51) | 678 (221) | 343 (277)

OUTCOME MEASURES:

1. Primary Outcome: Acromegaly Quality of Life (ACROQoL) Global Score
Description: The Global Score of the Acromegaly Quality of Life (ACROQoL) Survey measures quality of life in patients with acromegaly. Higher scores indicate better QOL. The range is 22-110 units on a scale.
Time Frame: Cross-sectional at baseline
Population: Patients receiving either no treatment (active acromegaly), pegvisomant monotherapy or somatostatin analog monotherapy from own doctor to treat acromegaly.
Measure: Mean (Standard Deviation); unit: points on a scale
Groups:
- Acromegaly With Pegvisomant; Acromegaly With Somatostatin Analog; Active Acromegaly: No adverse events were experienced in this study.
Arm/Group | Acromegaly With Pegvisomant | Acromegaly With Somatostatin Analog | Active Acromegaly
Number analyzed (Participants) | 29 | 55 | 32
points on a scale | 57 (19) | 60 (21) | 54 (22)

2. Secondary Outcome: The Gastrointestinal Quality of Life Index (GIQLI) Total Score
Description: The total score for the Gastrointestinal Quality of Life Index (GIQLI) measures quality of life with specific attention to gastrointestinal symptoms. The score ranges from 0-144 points on a scale. Higher scores indicating better quality of life.
Time Frame: Cross-sectional at baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Acomegaly With Pegvisomant | Acromegaly With Somatostatin Analog | Active Acromegaly
Number analyzed (Participants) | 29 | 55 | 32
points on a scale | 100 (21) | 107 (24) | 102 (22)

3. Secondary Outcome: 36-Item Short Form Survey Instrument (SF-36) Physical Health
Description: The Physical Health Summary Score of the SF-36 is a quality of life measure of physical health. It ranges from 0 to 100 points on a scale. Higher scores indicate better quality of life. This survey is scored as demonstrated at https://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html. The Physical Health Summary Score (Physical Component Summary) is calculated as the mean average of the physically relevant questions.
Time Frame: Cross-sectional at baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Groups:
- Acromegaly With Pegvisomant: Patients receiving pegvisomant monotherapy from own doctor to treat acromegaly.
Arm/Group | Acromegaly With Pegvisomant | Acromegaly With Somatostatin Analog | Active Acromegaly
Number analyzed (Participants) | 29 | 55 | 32
points on a scale | 60 (28) | 64 (28) | 63 (25)

4. Secondary Outcome: 36-Item Short Form Survey (SF-36) Mental Health Summary Score
Description: The Mental Health Summary Score of the SF-36 measures quality of life with a focus on mental health. It ranges from 0 to 100 points on a scale. Higher scores indicate better quality of life. This survey is scored as demonstrated at https://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html. The Mental Health Summary Score (Mental Component Summary) is calculated as the mean average of the emotionally relevant questions.
Time Frame: Cross-sectional at baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Acromegaly With Pegvisomant | Acromegaly With Somatostatin Analog | Active Acromegaly
Number analyzed (Participants) | 29 | 55 | 32
points on a scale | 58 (23) | 64 (25) | 58 (26)

ADVERSE EVENTS:
Time Frame: This was a cross-sectional study. Adverse events were collected at the baseline cross-sectional visit for each subject.
Groups:
- Acromegaly on Pegvisomant: Patients receiving pegvisomant monotherapy from own doctor to treat acromegaly.
- Acromegaly on Somatostatin Analog: Patients receiving somatostatin analog monotherapy from own doctor to treat acromegaly.
- Active Acromegaly: Patients receiving no medications to treat active acromegaly.
Arm/Group | Acromegaly on Pegvisomant | Acromegaly on Somatostatin Analog | Active Acromegaly
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/60 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/60 | 0/35
Other Adverse Events (participants affected / at risk) | 0/31 | 0/60 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No